CLINICAL TRIAL: NCT02587923
Title: A Retrospective Study on Safety, Diagnostic Yield and Therapeutic Effects of Endoscopic Unroofing for Small Gastric Subepithelial Tumors
Brief Title: Endoscopic Unroofing for Small Gastric SETs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Assistant Doctor, Medical University of Vienna
Other Study IDs: EK 1707/2015
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Small Gastric Subepithelial Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
Background: Accurate diagnosis of small gastric subepithelial tumors (SETs) is essential in order to assess their malignant potential. Endoscopic unroofing by conventional snare or needle knife has been reported to yield sufficient tissue samples for histological evaluation including immunohistochemical staining.

Aims: The investigators aim to evaluate endoscopic unroofing in patients with small gastric SETs regarding its safety and diagnostic accuracy as well as a potential therapeutic effect of this technique over time.

Methods: In the context of a retrospective analysis, the investigators will identify patients who underwent endoscopic unroofing of small SETs of the stomach at the Medical University of Vienna. Demographic data, indication for intervention, safety of the procedure and follow-up will be assessed.

DETAILED DESCRIPTION:
INTRODUCTION

Small gastric subepithelial tumors (SETs) are often incidental findings at upper endoscopy. Differential diagnoses include a variety of different pathologies such as gastrointestinal stromal tumors (GISTs), leiomyomas, leiomyosarcomas, lipomas, carcinoid tumors, granular cell tumors, duplication cysts or pancreatic rests. Since some of these entities have a potential of malignancy, accurate classification of gastric SETs is essential to define the best diagnostic and therapeutic management. Endosonography (EUS) is the current gold standard for further characterization of small gastric SETs. It provides differentiation between extra- and intramural lesions, information on the involvement of certain wall layers, measurement of a lesion as well as structural analysis according to the echogenicity of a lesion. Nevertheless, a level of uncertainty remains, even if a lesion shows a typical echo-pattern and layer involvement.

According to current guidelines, lesions of more than two centimeters in size that are suspected to be GISTs should be removed by surgical resection. Lesions less than one centimeter can be followed by annual EUS. For lesions bigger than one centimeter but smaller than two centimeters tissue sampling is recommended in order to correctly diagnose a lesion according to immunohistochemical markers (such as CD117 or CD34 in GISTs) and to quantify the malignant potential according to other histological factors (such as the mitotic index in GISTs) [1].

Tissue sampling can be done by using standard or jumbo forceps biopsy and EUS-guided fine needle aspiration or biopsy, but the diagnostic yield of these methods is rather low [2,3]. Better results can be achieved by endoscopic resection techniques such as endoscopic submucosal dissection (ESD), submucosal tunneling endoscopic resection or full thickness endoscopic resection [4,5]. The main advantage of these approaches is that they are not only diagnostic but also therapeutic strategies since the respective lesion can be resected as a whole comparable with conventional surgery. However, there is a high risk of procedure related adverse events such as bleeding or perforation (the latter is often unavoidable considering that most SETs are arising from deep wall layers such as the muscularis propria layer).

Endoscopic unroofing is very similar to the mentioned endoscopic resection techniques with the main difference that only partial resection is intended in order to get a representative tissue specimen for histological evaluation. This method has been described in a case series by Lee et al. in 2010 where it showed a very favorable diagnostic yield in gastric SETs [6]. To date, no study has reported on the follow-up of lesions investigated by endoscopic unroofing.

The aim of the present study is to evaluate endoscopic unroofing for small gastric SETs regarding safety, diagnostic yield and potential therapeutic effects over time.

PRIMARY HYPOTHESIS

Endoscopic unroofing has a high diagnostic accuracy in small gastric subepithelial tumors.

METHODS

This retrospective study will be conducted at the Division of Gastroenterology and Hepatology, Department of Internal Medicine III. Of the Medical University of Vienna. Patients who underwent endoscopic unroofing of gastric subepithelial tumors between 2000 and 2015 will be identified by searching the endoscopy reporting database "DOKMON". Clinical data will be collected from patients identified by reviewing endoscopy examination reports as well as other clinical documents including discharge letters in the report archiving database "AKIM". The following parameters will be assessed: Demographics (age, sex), indication for endoscopic unroofing, intraprocedural adverse events, hospital stay, histological result, follow-up procedures (including endoscopic or imaging controls, surgical resection). At the end of the study the mentioned parameters will be presented using descriptive statistics. Data analysis will be performed using SPSS 23.0. All patient related data will be de-identified using pseudonymization prior to any further processing.

SAMPLE SIZE

The investigators expect to encounter approximately 20 patients into this study (between 2000 and 2015).

ELIGIBILITY:
Inclusion criteria:

-) subjects with small gastric subepithelial tumors who underwent endoscopic unroofing

Exclusion criteria:

-) none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective series of patients treated at a tertiary university based center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Peri-interventional adverse events whether related or not
Diagnostic yield | 1 week
  Proportion of study patients with a histologically confirmed diagnosis after endoscopic unroofing.
Tumor status after endoscopic unroofing | 12 months
  Local result during follow up after endoscopic unroofing (proportion of patients with no change vs. partial remission vs. complete remission)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Dolak, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Background] Iorio N, Sawaya RA, Friedenberg FK. Review article: the biology, diagnosis and management of gastrointestinal stromal tumours. Aliment Pharmacol Ther. 2014 Jun;39(12):1376-86. doi: 10.1111/apt.12761. Epub 2014 Apr 20. PMID 24749828
- [Background] Buscaglia JM, Nagula S, Jayaraman V, Robbins DH, Vadada D, Gross SA, DiMaio CJ, Pais S, Patel K, Sejpal DV, Kim MK. Diagnostic yield and safety of jumbo biopsy forceps in patients with subepithelial lesions of the upper and lower GI tract. Gastrointest Endosc. 2012 Jun;75(6):1147-52. doi: 10.1016/j.gie.2012.01.032. Epub 2012 Mar 15. PMID 22425270
- [Background] Watson RR, Binmoeller KF, Hamerski CM, Shergill AK, Shaw RE, Jaffee IM, Stewart L, Shah JN. Yield and performance characteristics of endoscopic ultrasound-guided fine needle aspiration for diagnosing upper GI tract stromal tumors. Dig Dis Sci. 2011 Jun;56(6):1757-62. doi: 10.1007/s10620-011-1646-6. Epub 2011 Mar 1. PMID 21360279
- [Background] Zhou PH, Yao LQ, Qin XY, Cai MY, Xu MD, Zhong YS, Chen WF, Zhang YQ, Qin WZ, Hu JW, Liu JZ. Endoscopic full-thickness resection without laparoscopic assistance for gastric submucosal tumors originated from the muscularis propria. Surg Endosc. 2011 Sep;25(9):2926-31. doi: 10.1007/s00464-011-1644-y. Epub 2011 Mar 18. PMID 21424195
- [Background] Wilhelm D, von Delius S, Burian M, Schneider A, Frimberger E, Meining A, Feussner H. Simultaneous use of laparoscopy and endoscopy for minimally invasive resection of gastric subepithelial masses - analysis of 93 interventions. World J Surg. 2008 Jun;32(6):1021-8. doi: 10.1007/s00268-008-9492-1. PMID 18338207
- [Background] Lee CK, Chung IK, Lee SH, Lee SH, Lee TH, Park SH, Kim HS, Kim SJ, Cho HD. Endoscopic partial resection with the unroofing technique for reliable tissue diagnosis of upper GI subepithelial tumors originating from the muscularis propria on EUS (with video). Gastrointest Endosc. 2010 Jan;71(1):188-94. doi: 10.1016/j.gie.2009.07.029. Epub 2009 Oct 30. PMID 19879567
- [Derived] Dolak W, Beer A, Kristo I, Tribl B, Asari R, Schoniger-Hekele M, Wrba F, Schoppmann SF, Trauner M, Puspok A. A retrospective study on the safety, diagnostic yield, and therapeutic effects of endoscopic unroofing for small gastric subepithelial tumors. Gastrointest Endosc. 2016 Dec;84(6):924-929. doi: 10.1016/j.gie.2016.04.019. Epub 2016 Apr 22. PMID 27109457